CLINICAL TRIAL: NCT01527006
Title: An Open-label Pilot Study With an Extension Phase to Evaluate the Pharmacokinetics, and to Generate Preliminary Safety, Tolerability, and Efficacy of Perampanel (E2007) Oral Suspension When Given as an Adjunctive Therapy in Pediatric Subjects From 2 to Less Than 12 Years of Age With Epilepsy
Brief Title: Pharmacokinetics, Efficacy, and Safety of Perampanel Oral Suspension on Seizure Frequency in Pediatric Subjects Maintained on One to Three Stable Antiepileptic Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-G000-232
Record Dates: First submitted 2011-11-10; First posted 2012-02-06 (Estimated); Results first posted 2015-08-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Central Nervous System
MeSH Terms: interventions — perampanel

ARMS (1):
- perampanel (Experimental): Age Cohort 1 ( greater than or equal to 7 to less than 12 years of age at time of consent/assent) and age Cohort 2 ( greater than or equal to 2 to less than 7 years of age).
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — During the titration period, participants started at a set daily dose of 0.015 mg/kg and had doses up-titrated at 1-week intervals (6 titration steps) to a maximum daily dose of 0.18 mg/kg. During the Maintenance Period, participants continued taking perampanel oral suspension once daily at the dose level they achieved at the end of the Titration Period. During the extension phase, participants continued taking perampanel oral suspension once daily, at the dose level achieved at the end of the treatment phase of the core study to a maximum daily dose of 0.18 mg/kg. The maximum total daily dose a participant was allowed was 12 mg.

SUMMARY:
This study is designed to evaluate the pharmacokinetics, efficacy, and safety of perampanel oral suspension on seizure frequency in pediatric participants maintained on one to three stable antiepileptic drugs

DETAILED DESCRIPTION:
This is a multicenter, multiple ascending dose, open-label study (Core Study) with an Extension Phase. The Core Study consisted of 2 phases, the Pretreatment Phase and the Treatment Phase. The Pretreatment Phase lasted up to 2 weeks in duration, during which participants were assessed for their eligibility to participate in the study. The Treatment Phase consisted of 3 periods: Titration (7 weeks), Maintenance (4 weeks), and Follow-up (4 weeks; only for those participants not rolling over into the Extension Phase after completing the Treatment Phase and for those participants who discontinued from the study). All subjects who completed all scheduled visits up to and including the final visit of the Treatment Phase (Core Study) were eligible to participate in the Extension Phase of the study. The Extension Phase consisted of 2 periods: Maintenance (41 weeks) and Follow-up (4 weeks).

ELIGIBILITY:
Inclusion:

1. Have a minimum weight of 10 kg (22 lb)
2. Have had brain imaging (computed tomography [CT] or magnetic resonance imaging [MRI]) prior to Visit 1 that ruled out a progressive cause of epilepsy
3. Have a diagnosis of epilepsy with any type of seizure according to the International League Against Epilepsy's (ILAE) Classification of Epileptic Seizures (1981). Diagnosis should have been established at least 6 months prior to Visit 1, by clinical history and an electroencephalogram (EEG) that is consistent with epilepsy; normal interictal EEGs will be allowed provided that the participant meets the other diagnosis criterion (i.e. clinical history)
4. Have had one or more seizure(s) during the 4 weeks prior to Visit 1
5. Are currently being treated with stable doses of one to a maximum of three AEDs for at least 4 weeks prior to Visit 1 and throughout the study duration (Only one perampanel inducing AED [i.e. carbamazepine, oxcarbazepine, phenytoin] out of the maximum of 3 AEDs is allowed in at least one third of the participants in each age cohort and not to exceed one half of the population of each age cohort. The remaining participants should not be taking any inducer)
6. Have been on their current concomitant AED regimen for 2 months or more with a stable dose for at least 4 weeks prior to Visit 1
7. Must have discontinued all restricted medications at least 2 weeks or five half-lives (whichever is longer) prior to Visit 1
8. Females aged at least 8 years or of child-bearing potential must have a negative serum beta-hCG at Visit 1 and a negative urine pregnancy test prior to titration at Visit 2. Female participants of childbearing potential must agree for the duration of the study and for a period of at least 60 days following administration of the last dose of study drug to be abstinent or commit to the consistent and correct use of a medically acceptable method of birth control (e.g., a double-barrier method [condom + spermicide, condom + diaphragm with spermicide])

Exclusion:

1. Have a history of status epilepticus that required hospitalization during the 6 months prior to Visit 1
2. Have current or a history of pseudo-seizures (psychogenic non-epileptic seizures [PNES]) from birth or within approximately 5 years prior to Visit 1
3. Have seizures due to treatable medical conditions, such as those arising due to metabolic disturbances, toxic exposure, or an active infection
4. Have epilepsy secondary to progressive cerebral disease or any other progressive neurodegenerative disease
5. Have had epilepsy surgery within 1 year prior to Visit 1
6. Are scheduled and/or confirmed to have epilepsy surgery within 6 months after Visit 1; however, those who have previously documented failed epilepsy surgery will be allowed
7. Use of intermittent rescue benzodiazepines (i.e. 1-2 doses over a 24-hour period considered one-time rescue) two or more times in a 30-day period prior to Visit 1
8. If felbamate is used as a concomitant AED, participants must be on felbamate for at least 2 years, with a stable dose for 8 weeks prior to Visit 1. They must not have a history of white blood cell (WBC) count below 2500/L (2.50 x 10^9/L), platelets below 100,000, liver function tests (LFTs) above 3 times the upper limit of normal (ULN), or other indication of hepatic or bone marrow dysfunction while receiving felbamate. If participants received felbamate in the past, it must have been discontinued 8 weeks prior to Visit 1
9. Have concomitant use of vigabatrin: participants who took vigabatrin in the past must be off vigabatrin for approximately 5 months prior to Visit 1 and must have documentation showing no evidence of a vigabatrin-associated clinically significant abnormality in the visual perimetry test
10. If ketogenic diet is used, participants must be on a stable regimen for at least 4 weeks prior to Visit 1
11. Have previously participated in a clinical trial involving perampanel

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 63 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Gee, Study Director — Eisai Limited
Locations (23):
- United States (23):
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Gulf Breeze, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Augusta, Georgia
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Shreveport, Louisiana
  - Chesterfield, Missouri
  - Columbia, Missouri
  - Gibbsboro, New Jersey
  - Buffalo, New York
  - Akron, Ohio
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Richmond, Virginia

REFERENCES:
- [Derived] Renfroe JB, Mintz M, Davis R, Ferreira J, Dispoto S, Ferry J, Umetsu Y, Rege B, Majid O, Hussein Z, Laurenza A. Adjunctive Perampanel Oral Suspension in Pediatric Patients From >/=2 to <12 Years of Age With Epilepsy: Pharmacokinetics, Safety, Tolerability, and Efficacy. J Child Neurol. 2019 Apr;34(5):284-294. doi: 10.1177/0883073819827407. Epub 2019 Feb 10. PMID 30739576

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 63 participants who were enrolled, 13 participants were screen failures and 50 participants were eligible to continue in the Core Study. Of the 42 subjects who completed the Core Study, 41 subjects continued into the Extension Phase.
Groups:
- Cohort ( ≥ 2 to < 7 Years of Age); Cohort ( ≥ 7 to < 12 Years of Age): During the titration period, participants started at a set daily dose of 0.015 mg/kg and had doses up-titrated at 1-week intervals (6 titration steps) to a maximum daily dose of 0.18 mg/kg. During the Maintenance Period, participants continued taking perampanel oral suspension once daily at the dose level they achieved at the end of the Titration Period. During the extension phase, participants continued taking perampanel oral suspension once daily, at the dose level achieved at the end of the treatment phase of the core study to a maximum daily dose of 0.18 mg/kg. The maximum total daily dose a participant was allowed was 12 mg.
Period: Core Study
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) | Cohort ( ≥ 7 to < 12 Years of Age)
Started | 22 | 28
Completed | 20 | 22
Not Completed | 2 | 6
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject Choice | 1 | 0
Not completed — Inadequate Therapeutic Effect | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other | 0 | 2
Period: Extension Phase
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) | Cohort ( ≥ 7 to < 12 Years of Age)
Started | 19 (Of the 20 subjects who completed the Core Study, 19 subjects continued into the Extension Phase.) | 22
Completed | 13 | 14
Not Completed | 6 | 8
Not completed — Adverse Event | 4 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Subject Choice | 1 | 1
Not completed — Inadequate therapeutic effect | 1 | 1
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study; Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study: During the titration period, participants started at a set daily dose of 0.015 mg/kg and had doses up-titrated at 1-week intervals (6 titration steps) to a maximum daily dose of 0.18 mg/kg. During the Maintenance Period, participants continued taking perampanel oral suspension once daily at the dose level they achieved at the end of the Titration Period.
- Total: Total of all reporting groups
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study | Total
Number analyzed (Participants) | 22 | 28 | 50
Age, Continuous [Median (Full Range); unit: Years] | 5 [2 to 6] | 9 [7 to 11] | 7.5 [2 to 11]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 15 | 19 | 34

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline in Seizure Frequency Per 28 Days in Treatment Phase [Core Study]
Description: Seizure frequency was derived from information (seizure count and type) recorded in participant diary. The seizure frequency per 28 days was calculated the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. The percent change in 28-day seizure frequency from baseline was assessed for overall seizures, overall partial seizures, overall generalized seizures, and unclassified seizures. The data is presented as mean percent change +/- standard deviation.
Time Frame: Baseline [2 weeks Pretreatment Phase (Visit 1) plus 4 weeks Prior to Pretreatment Phase], Week 0 to Week 15
Population: The full analysis set, defined as participants who received study drug, had any seizure frequency data during the 2-week Pretreatment Phase plus the 4 weeks prior to the Pretreatment Phase (Visit 1), and during the Treatment Phase of the Core Study.
Measure: Median (Full Range); unit: Percent change
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 22 | 28
Percent change
  Overall seizures | -43.6 [-100 to 95.4] | -33.9 [-100 to 1038.9]
  Overall partial seizures | -82.5 [-100 to 95.4] | -46.8 [-100 to 1722.2]
  Overall generalized seizures | -53.1 [-100 to 188.7] | 305.4 [-62.9 to 1277.3]
  Unclassified Seizures | -73.7 [-100 to 217.3] | -67.3 [-100 to -34.6]

2. Primary Outcome: Apparent Clearance (CL/F) of Perampanel [Core Study]
Description: CL/F was defined as the volume of plasma cleared of the drug per unit time. Blood samples were collected at day 8, Day 36, Day 64 , and Day 78. The CL/F values were calculated for each visit and averaged to derive the total CL/F value per arm. Data was analyzed for 2 categories: CYP3A4/5 inducers (carbamazepine, oxcarbazepine and phenytoin) and non-inducers. Data is presented as mean Liter per hour +/-standard deviation.
Time Frame: From Day 8 up to Day 78
Population: The pharmacokinetic (PK) analysis set, defined as participants with at least 1 pharmacokinetic assessment of perampanel with a documented dosing history.
Measure: Mean (Standard Deviation); unit: Liter per hour
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 20 | 22
Liter per hour
  Non-Inducers (N=14, 12) | 0.732 (0.374) | 0.956 (0.4)
  Inducers (N=6, 10) | 1.73 (1.18) | 1.92 (0.517)

3. Secondary Outcome: 50% Responder Rate During the Maintenance Period-LOCF [Core Study]
Description: Responder rate was defined as the proportion of participants with a 50% decrease in 28-day seizure frequency during the Maintenance Period compared to Baseline [2 weeks Pretreatment Phase (Visit 1) plus 4 Weeks Prior to Pretreatment Phase] for overall seizures, overall partial seizures, overall generalized seizures, and unclassified seizures. The data is presented as percent responders. LOCF = Last Observation Carried Forward.
Time Frame: Baseline [2 weeks Pretreatment Phase (Visit 1) plus 4 weeks Prior to Pretreatment Phase], Week 9 to 11
Population: as for outcome 1
Measure: Number; unit: Percent responders
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 22 | 28
Percent responders
  Overall seizures | 72.7 | 53.8
  Overall partial seizures | 82.4 | 60.9
  Overall generalized seizures | 76.9 | 33.3
  Unclassified Seizures | 66.7 | 100

4. Secondary Outcome: Seizure-free Rate During the Maintenance Period [Core Study]
Description: Seizure-free rate, defined as the percentage of participants who were seizure-free during the Maintenance Period. SG = Secondary Generalization.
Time Frame: Week 9 to Week 11
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 20 | 22
Percentage of participants
  Overall Seizures | 15 | 27.3
  Simple Partial without Motor Signs | 100 | 100
  Simple Partial with Motor signs | 80 | 95.5
  Complex Partial | 80 | 50
  Partial Seizures with SG | 75 | 90.9
  Overall Partial Seizures | 50 | 45.5
  Absence Generalized | 95 | 90.9
  Myoclonic Generalized | 80 | 86.4
  Clonic Generalized | 100 | 100
  Tonic Generalized | 85 | 90.9
  Tonic Clonic Generalized | 80 | 90.9
  Atonic Generalized | 95 | 95.5
  Overall Generalized seizures | 55 | 77.3
  Unclassified Seizures | 100 | 95.5

5. Secondary Outcome: The Clinical Global Impression of Change at the End of Treatment (EOT) [Core Study]
Description: The Clinical Global Impression (CGI) evaluated perceived seizure frequency and severity, the occurrence of AEs, and overall functional status of the participant. The investigator performed the Clinical Global Impression of Severity for all participants at Baseline (Week 0). The evaluation used a 7-point scale where 1=normal, not at all ill and 7=extremely ill. The investigator performed the Clinical Global Impression of Change for all participants at the EOT (the duration after the day of first study drug dose up to 7 days after the last Core Phase drug dose, inclusive). The evaluation used a 7-point scale where 1=very much improved and 7=very much worse. This tool was used to assess the participant's status over the 4-week period prior to its completion compared to Baseline (Week 0).
Time Frame: Week 0 (Baseline), Week 11 or EOT
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 22 | 27
Participants
  Baseline - Normal, not at all ill (N=22, 27) | 6 | 5
  Baseline - Borderline mentally ill (N=22, 27) | 0 | 0
  Baseline - Mildly ill (N=22, 27) | 3 | 4
  Baseline - Moderately ill (N=22,27) | 10 | 11
  Baseline - Markedly ill (N=22, 27) | 3 | 4
  Baseline - Severely ill (N=22, 27) | 0 | 3
  Baseline - Extremely ill (N=22, 27) | 0 | 0
  EOT - Very much improved (N=22, 25) | 6 | 7
  EOT - Much improved (N=22, 25) | 8 | 8
  EOT - Minimally improved (N=22, 25) | 5 | 5
  EOT - No Change (N=22, 25) | 2 | 3
  EOT - Minimally worse (N=22, 25) | 0 | 1
  EOT - Much worse (N=22, 25) | 0 | 1
  EOT - Very much worse (N=22, 25) | 1 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Non-Serious Adverse Events (AEs) and Treatment Emergent Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Perampanel
Description: An AE was defined as any untoward medical occurrence in a participant administered with the study drug. A SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening (ie, the participant was at immediate risk of death from the AE as it occurred; this did not include an event that, had it occurred in a more severe form or was allowed to continue, might have caused death), required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was as a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). In this study, treatment emergent AEs (defined as an AE (serious/non-serious) that started/increased in severity on/after the first dose of study drug up to 30 days after the final dose of study drug) were assessed. The details of the adverse events are presented in the safety section of the results.
Time Frame: For each participant, from the first treatment dose till 30 days after the last dose or up to Week 15 for Core Study and Week 56 for the Extension Phase
Population: The Safety Analysis Set included all subjects who took at least 1 dose of perampanel and had at least 1 postdose safety assessment during the Core Study and the Extension Phase.
Measure: Number; unit: Participants
Groups:
- Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase; Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase: During the extension phase, participants continued taking perampanel oral suspension once daily, at the dose level achieved at the end of the treatment phase of the core study to a maximum daily dose of 0.18 mg/kg. The maximum total daily dose a participant was allowed was 12 mg.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Number analyzed (Participants) | 22 | 28 | 19 | 22
Participants
  Treatment Emergent Non-Serious AEs | 22 | 25 | 19 | 22
  Treatment Emergent SAEs | 3 | 5 | 6 | 7

7. Secondary Outcome: Palatability Questionnaire Assessment - How Does This Medicine Taste [Core Study]
Description: The Palatability Questionnaire was answered directly by participants in Cohort ( ≥ 7 to ≤ 12 years) and indirectly by participants in Cohort ( ≥ 2 to ≤ 7 years) via their parents/caregivers. Participants selected their response from one of the five options (very good, good, not good-not bad, bad, very bad).
Time Frame: Week 5 or at the time of early discontinuation
Population: The Safety Analysis Set, defined as participants who received study drug treatment and had at least 1 postdose safety assessment.
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 13 | 19
Participants
  Very good | 3 | 3
  Good | 6 | 7
  Not good, not bad | 2 | 3
  Bad | 2 | 3
  Very bad | 0 | 3

8. Secondary Outcome: Palatability Questionnaire Assessment - How Does This Medicine Smell [Core Study]
Description: as for outcome 7
Time Frame: Week 5 or at the time of early discontinuation
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 13 | 19
Participants
  Very good | 0 | 2
  Good | 5 | 3
  Not good, not bad | 7 | 13
  Bad | 1 | 0
  Very bad | 0 | 1

9. Secondary Outcome: Palatability Questionnaire Assessment - Based on Its Taste, Smell, and How it Felt in the Mouth, How Easy or Difficult Was it for You / Your Child to Take This Medicine Every Day [Core Study]
Description: The Palatability Questionnaire was answered directly by participants in Cohort ( ≥ 7 to ≤ 12 years) and indirectly by participants in Cohort ( ≥ 2 to ≤ 7 years) via their parents/caregivers. Participants selected their response from one of the five options (very easy, easy, neither easy or difficult, difficult and very difficult).
Time Frame: Week 5 or at the time of early discontinuation
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 14 | 19
Participants
  Very easy | 6 | 7
  Easy | 5 | 7
  Neither easy or difficult | 3 | 3
  Difficult | 0 | 1
  Very Difficult | 0 | 1

10. Primary Outcome: Steady-state Average Concentration (C av,ss) of Perampanel [Core Study]
Description: C av,ss was calculated as 'Dose (mg)/Dosing Interval (24 h)/(CL/F [L/h]) x 1000'. C av,ss during a dosing interval was dose-normalized to 0.12 mg/kg in participants aged ≥ 2 to less than 12 years (intended to correspond to 8 mg/70 kg in adults/adolescents). Blood samples were collected at day 8, Day 36, Day 64 , and Day 78. C av,ss values were calculated for each visit and averaged to derive the total C av,ss value per arm. Data was analysed for 2 categories: CYP3A4/5 inducers (carbamazepine, oxcarbazepine and phenytoin) and non-inducers. Data is presented as mean Liter per hour +/- standard deviation.
Time Frame: From Day 8 up to Day 78
Population: The PK analysis set, defined as participants with at least 1 pharmacokinetic assessment of perampanel with a documented dosing history.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 20 | 22
ng/mL
  Non-Inducers (N=14, 12) | 179 (110) | 266 (220)
  Inducers (N=6, 10) | 96.8 (90.4) | 105 (38.9)

11. Secondary Outcome: Palatability Questionnaire Assessment - Would You/Your Child Have Preferred This Medicine to Have Been Flavored, e.g. Fruity [Core Study]
Description: The Palatability Questionnaire was answered directly by participants in Cohort ( ≥ 7 to ≤ 12 years) and indirectly by participants in Cohort ( ≥ 2 to ≤ 7 years) via their parents/caregivers. Participants selected their response from one of the three options (yes, no and don't mind).
Time Frame: Week 5 or at the time of early discontinuation
Population: as for outcome 7
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 15 | 19
Participants
  Yes | 4 | 9
  No | 2 | 5
  Don't mind | 9 | 5

12. Other Pre Specified Outcome: The Effect of Demographics on Population PK Parameters: AUC
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: The Effect of Demographics on Population PK Parameters: Cmax
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

14. Other Pre Specified Outcome: The Effect of Demographics on Population PK Parameters: Tmax
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

15. Other Pre Specified Outcome: The Effect of the Most Common Concomitant AEDs on Population PK Parameters: AUC
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

16. Other Pre Specified Outcome: The Effect of the Most Common Concomitant AEDs on Population PK Parameters: Cmax
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

17. Other Pre Specified Outcome: The Effect of the Most Common Concomitant AEDs on Population PK Parameters: Tmax
Description: This outcome was not assessed in the study.
Time Frame: 11 weeks
Population: This outcome was not assessed in the study.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Percentage Change From Baseline in Seizure Frequency Per 28 Days During the Overall Treatment Duration by 13-week Intervals [Extension Phase]
Description: as for outcome 1
Time Frame: Baseline [2 weeks Pretreatment Phase (Visit 1) plus 4 weeks Prior to Pretreatment Phase], Weeks 1-13, Weeks 14-26, Weeks 27-39, and Weeks 40-52
Population: The Full Analysis Set included all subjects who took at least 1 dose of perampanel during the Extension Phase, and had any seizure frequency data during the 2-week Pretreatment Phase plus the 4 weeks prior to Pretreatment Phase (Visit 1) of the Core Study and had any seizure frequency data during the Extension Phase.
Measure: Median (Full Range); unit: Percent change
Groups:
- Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase; Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase: During the titration period, participants started at a set daily dose of 0.015 mg/kg and had doses up-titrated at 1-week intervals (6 titration steps) to a maximum daily dose of 0.18 mg/kg. During the Maintenance Period, participants continued taking perampanel oral suspension once daily at the dose level they achieved at the end of the Titration Period. During the extension phase, participants continued taking perampanel oral suspension once daily, at the dose level achieved at the end of the treatment phase of the core study to a maximum daily dose of 0.18 mg/kg. The maximum total daily dose a participant was allowed was 12 mg.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Number analyzed (Participants) | 19 | 22
Percent change
  Overall Seizures- Weeks 1-13 | -58.74 [-100.0 to 75.8] | -39.59 [-100.0 to 759.3]
  Overall Seizures- Weeks 14-26 | -76.89 [-100.0 to 134.4] | -39.19 [-100.0 to 389.8]
  Overall Seizures- Weeks 27-39; N=18, 20 | -80.93 [-100.0 to 129.9] | -45.60 [-100.0 to 474.6]
  Overall Seizures- Weeks 40-52; N=15, 15 | -77.58 [-100.0 to -1.2] | -47.25 [-100.0 to 200.0]
  Overall Partial Seizures- Weeks 1-13; N=14,19 | -79.62 [-100.0 to 75.8] | -56.04 [-100.0 to 290.5]
  Overall Partial Seizures- Weeks 14-26; N=14, 19 | -78.69 [-100.0 to 134.4] | -67.30 [-100.0 to 87.9]
  Overall Partial Seizures- Weeks 27-39; N=14, 17 | -89.49 [-100.0 to 129.9] | -53.57 [-100.0 to 165.2]
  Overall Partial Seizures- Weeks 40-52; N=14, 14 | -89.89 [-100.0 to -1.2] | -39.46 [-100.0 to 100.0]
  Overall Generalized Seizures- Weeks 1-13; N=11, 6 | -63.96 [-100.0 to 465.5] | 177.58 [-65.0 to 1065.4]
  Overall Generalized Seizures- Weeks 14-26; N=11, 6 | -79.08 [-100.0 to 440.7] | -14.13 [-87.3 to 389.8]
  Overall Generalized Seizures- Weeks 27-39; N=10, 6 | -73.93 [-100.0 to -8.9] | -4.77 [-83.6 to 474.6]
  Overall Generalized Seizures- Weeks 40-52; N=7, 3 | -76.91 [-100.0 to 182.8] | -5.86 [-61.5 to 700.0]
  Unclassified Epileptic Seizure- Weeks 1-13; N=2, 1 | -88.74 [-100.0 to 77.5] | -41.61 [-41.61 to -41.61]
  Unclassified Epileptic Seizure- Weeks 14-26; N=2,1 | -100.0 [-100.0 to -100.0] | -21.07 [-21.07 to -21.07]
  Unclassified Epileptic Seizure- Weeks 27-39; N=2,1 | -58.24 [-100.0 to -16.5] | 6.81 [6.81 to 6.81]
  Unclassified Epileptic Seizure- Weeks 40-52; N=2,1 | -100.0 [-100.0 to -100.0] | -73.21 [-73.21 to -73.21]

19. Secondary Outcome: 50 % Responder Rate During the Overall Treatment Duration by 13-week Intervals [Extension Phase]
Description: Responder rate was defined as the proportion of participants with a 50% decrease in 28-day seizure frequency during the overall treatment duration. The percentage of responders was assessed from Week 1 of perampanel treatment through successive 13-week intervals for overall seizures, overall partial seizures, overall generalized seizures, and unclassified seizures with baseline as Pretreatment Phase (Visit 1) of 2 weeks plus 4 weeks Prior to Pretreatment Phase. The data is presented as percentage of responders.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: Percentage of responders
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Number analyzed (Participants) | 19 | 22
Percentage of responders
  Overall Seizures- Weeks 1-13 | 57.9 | 45.5
  Overall Seizures- Weeks 14-26 | 84.2 | 45.5
  Overall Seizures- Weeks 27-39; N=18, 20 | 77.8 | 45.0
  Overall Seizures- Weeks 40-52; N=15, 15 | 80.0 | 46.7
  Overall Partial Seizures- Weeks 1-13; N=14,19 | 64.3 | 57.9
  Overall Partial Seizures- Weeks 14-26; N=14, 19 | 85.7 | 57.9
  Overall Partial Seizures- Weeks 27-39; N=14, 17 | 92.9 | 52.9
  Overall Partial Seizures- Weeks 40-52; N=14, 14 | 71.4 | 42.9
  Overall Generalized Seizures- Weeks 1-13; N=11, 6 | 72.7 | 16.7
  Overall Generalized Seizures- Weeks 14-26; N=11, 6 | 81.8 | 33.3
  Overall Generalized Seizures- Weeks 27-39; N=10, 6 | 70.0 | 16.7
  Overall Generalized Seizures- Weeks 40-52; N=7, 3 | 71.4 | 33.3
  Unclassified Epileptic Seizure- Weeks 1-13; N=2, 1 | 100.0 | 0.0
  Unclassified Epileptic Seizure- Weeks 14-26; N=2,1 | 100.0 | 0.0
  Unclassified Epileptic Seizure- Weeks 27-39; N=2,1 | 50.0 | 0.0
  Unclassified Epileptic Seizure- Weeks 40-52; N=2,1 | 100.0 | 100.0

20. Secondary Outcome: Seizure-free Rate During the Overall Treatment Duration [Extension Phase]
Description: Seizure-free rate, defined as the percentage of participants who were seizure-free during the Maintenance Period. The percentage of participants who were seizure free was assessed from Week 1 of perampanel treatment through successive 13-week intervals for overall seizures, overall partial seizures, overall generalized seizures, and unclassified seizures with baseline as Pretreatment Phase (Visit 1) of 2 weeks plus 4 weeks Prior to Pretreatment Phase. The data is presented as the percentage of participants.
Time Frame: as for outcome 18
Population: as for outcome 18
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Number analyzed (Participants) | 19 | 22
Percentage of participants
  Overall Seizures- Weeks 1-13 | 21.1 | 22.7
  Overall Seizures- Weeks 14-26;N=18, 20 | 22.2 | 30.0
  Overall Seizures- Weeks 27-39; N=15, 15 | 13.3 | 33.3
  Overall Seizures- Weeks 40-52; N=11, 11 | 27.3 | 36.4
  Overall Partial Seizures- Weeks 1-13 | 52.6 | 40.9
  Overall Partial Seizures- Weeks 14-26; N=18, 20 | 55.6 | 45.0
  Overall Partial Seizures- Weeks 27-39; N=15, 15 | 33.3 | 40.0
  Overall Partial Seizures- Weeks 40-52; N=11, 11 | 36.4 | 45.5
  Overall Generalized Seizures- Weeks 1-13 | 57.9 | 72.7
  Overall Generalized Seizures- Weeks 14-26; N=18,20 | 55.6 | 75.0
  Overall Generalized Seizures- Weeks 27-39; N=15,15 | 66.7 | 80.0
  Overall Generalized Seizures- Weeks 40-52; N=11,11 | 63.6 | 90.9
  Unclassified Epileptic Seizure- Weeks 1-13 | 100.0 | 90.9
  Unclassified Epileptic Seizure-Weeks 14-26;N=18,20 | 100.0 | 95.0
  Unclassified Epileptic Seizure-Weeks 27-39;N=15,15 | 93.3 | 93.3
  Unclassified Epileptic Seizure-Weeks 40-52;N=11,11 | 100.0 | 90.9

21. Secondary Outcome: The Clinical Global Impression of Change During the Overall Treatment Duration by Visit and at EOT [Extension Phase]
Description: The Clinical Global Impression (CGI) evaluated perceived seizure frequency and severity, the occurrence of AEs, and overall functional status of the participant. The investigator performed the Clinical Global Impression of Severity for all participants at Baseline (Week 0). The evaluation used a 7-point scale where 1=normal, not at all ill and 7=extremely ill. The investigator performed the Clinical Global Impression of Change for all participants at planned visit and at EOT (the duration after the day of first study drug dose up to 7 days after the Extension Phase drug dose, inclusive). The evaluation used a 7-point scale where 1=very much improved and 7=very much worse. This tool was used to assess the participant's status over the 4-week period prior to the planned/EOT visits compared to Baseline (Week 0).
Time Frame: Week 0 (Baseline), Week 11, Week 28, Week 52 or EOT
Population: as for outcome 18
Measure: Number; unit: Participants
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Number analyzed (Participants) | 19 | 22
Participants
  Baseline- Normal, not at all ill | 5 | 3
  Baseline- Borderline mentally ill | 0 | 0
  Baseline- Mildly ill | 3 | 4
  Baseline- Moderately ill | 10 | 10
  Baseline- Markedly ill | 1 | 4
  Baseline- Severely ill | 0 | 1
  Baseline- Extremely ill | 0 | 0
  Week 11- Very much improved; N=19, 21 | 6 | 7
  Week 11- Much improved; N=19, 21 | 8 | 7
  Week 11- Minimally improved; N=19, 21 | 3 | 5
  Week 11- No change; N= 19, 21 | 2 | 2
  Week 11- Minimally worse; N=19, 21 | 0 | 0
  Week 11- Much worse; N=19, 21 | 0 | 0
  Week 11- Very much worse; N=19, 21 | 0 | 0
  Week 28- Very much improved; N=18, 19 | 5 | 4
  Week 28- Much improved; N=18, 19 | 7 | 8
  Week 28- Minimally improved; N=18, 19 | 2 | 3
  Week 28- No change; N=18, 19 | 4 | 3
  Week 28- Minimally worse; N=18, 19 | 0 | 1
  Week 28- Much worse; N=18, 19 | 0 | 0
  Week 28- Very much worse; N=18, 19 | 0 | 0
  Week 52- Very much improved; N=14, 12 | 1 | 3
  Week 52- Much improved; N=14, 12 | 7 | 5
  Week 52- Minimally improved; N=14, 12 | 4 | 4
  Week 52- No change; N=14, 12 | 1 | 0
  Week 52- Minimally worse; N=14, 12 | 0 | 0
  Week 52- Much worse; N=14, 12 | 1 | 0
  Week 52- Very much worse; N=14, 12 | 0 | 0
  EOT- Very much improved | 1 | 4
  EOT- Much improved | 8 | 9
  EOT- Minimally improved | 5 | 6
  EOT- No change | 4 | 2
  EOT- Minimally worse | 0 | 1
  EOT- Much worse | 1 | 0
  EOT- Very much worse | 0 | 0

ADVERSE EVENTS:
Time Frame: For each participant, from the first treatment dose till 30 days after the last dose or up to Week 15 for Core Study and Week 56 for the Extension Phase
Description: Treatment emergent AEs are presented in this section. The Safety Analysis Set included all subjects who took at least 1 dose of perampanel and had at least 1 postdose safety assessment during the Core Study and the Extension Phase.
Arm/Group | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase
Serious Adverse Events (participants affected / at risk) | 3/22 | 5/28 | 6/19 | 7/22
Other Adverse Events (participants affected / at risk) | 22/22 | 25/28 | 19/19 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study (N=22) | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study (N=28) | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase (N=19) | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase (N=22)
Developmental Hip Dysplasia (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 1 | 0 | 1
Otitis Media Acute (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 0 | 1 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1 | 2 | 1
Abnormal Behaviour (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
Cyanosis (Cardiac disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cyclic Vomiting Syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 1 | 0
Anticonvulsant Drug Level Increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle Contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Status Epilepticus (Nervous system disorders) | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort ( ≥ 2 to < 7 Years of Age) - For Core Study (N=22) | Cohort ( ≥ 7 to < 12 Years of Age) - For Core Study (N=28) | Cohort ( ≥ 2 to < 7 Years of Age) - For Extension Phase (N=19) | Cohort ( ≥ 7 to < 12 Years of Age) - For Extension Phase (N=22)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 4 | 0 | 5
Vomiting (Gastrointestinal disorders) | 3 | 5 | 4 | 6
Fatigue (General disorders) | 1 | 8 | 1 | 6
Gait Disturbance (General disorders) | 2 | 1 | 2 | 0
Irritability (General disorders) | 3 | 5 | 3 | 5
Pyrexia (General disorders) | 8 | 4 | 8 | 7
Ear Infection (Infections and infestations) | 0 | 2 | 3 | 4
Otitis Media (Infections and infestations) | 2 | 2 | 2 | 3
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 2 | 5 | 6
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1
Thyroxine Decreased (Investigations) | 0 | 2 | 0 | 2
Weight Increased (Investigations) | 1 | 3 | 1 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 2 | 2 | 1
Increased Aappetite (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4
Ataxia (Nervous system disorders) | 0 | 2 | 0 | 2
Balance Disorder (Nervous system disorders) | 1 | 2 | 1 | 1
Dizziness (Nervous system disorders) | 3 | 2 | 3 | 2
Headache (Nervous system disorders) | 1 | 2 | 2 | 3
Lethargy (Nervous system disorders) | 1 | 2 | 4 | 3
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 2 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 3 | 3 | 3
Tremor (Nervous system disorders) | 0 | 2 | 0 | 0
Aggression (Psychiatric disorders) | 3 | 1 | 5 | 2
Anxiety (Psychiatric disorders) | 2 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 1 | 2
Oppositional Defiant Disorder (Psychiatric disorders) | 2 | 1 | 2 | 1
Tearfulness (Psychiatric disorders) | 2 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 1
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1
Eye Irritation (Eye disorders) | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Aphthous Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival Recession (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Oral Mucosal Discolouration (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Autoimmune Disorder (Immune system disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Atypical Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 2
Clostridium Difficile Infection (Infections and infestations) | 0 | 0 | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 1
Lice Infestation (Infections and infestations) | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 3 | 3
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Tinea Capitis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral Rash (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Epiphyseal Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Blood Bicarbonate Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Sodium Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Triglycerides Increased (Investigations) | 0 | 0 | 1 | 0
Blood Uric Acid Decreased (Investigations) | 0 | 0 | 2 | 1
Cardiac Murmur (Investigations) | 0 | 0 | 1 | 0
Cardiac Murmur Functional (Investigations) | 0 | 0 | 1 | 0
Globulins Decreased (Investigations) | 0 | 0 | 1 | 0
Heart Rate Increased (Investigations) | 0 | 0 | 1 | 0
Tri-Iodothyronine Decreased (Investigations) | 0 | 0 | 1 | 0
Weight Decreased (Investigations) | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Posture Abnormal (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 2 | 0
Drooling (Nervous system disorders) | 0 | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0
Intention Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0
Speech Disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal Behaviour (Psychiatric disorders) | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed Mood (Psychiatric disorders) | 0 | 0 | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 1 | 0
Echolalia (Psychiatric disorders) | 0 | 0 | 1 | 0
Emotional Disorder (Psychiatric disorders) | 0 | 0 | 2 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Mood Altered (Psychiatric disorders) | 0 | 0 | 1 | 0
Mood Swings (Psychiatric disorders) | 0 | 0 | 0 | 2
Sleep Disorder (Psychiatric disorders) | 0 | 0 | 2 | 1
Suicidal Ideation (Psychiatric disorders) | 0 | 0 | 1 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Enuresis (Renal and urinary disorders) | 0 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Vulval Disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Grunting (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other